CLINICAL TRIAL: NCT02784314
Title: Medico-economic Evaluation of Robotic-assisted Radical Prostatectomy Versus Laparoscopic Radical Prostatectomy
Brief Title: Cost Efficacy Evaluation of Robot Assisted Radical Prostatectomy
Acronym: ROBOTCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009.587
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
Keywords: Clinically localized prostate cancer; Robotic-assisted prostatectomy; Laparoscopic prostatectomy; Erectile function ;; Cost efficacy study
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic-Assisted Radical Prostatectomy (Experimental): Robotic-Assisted Radical Prostatectomy using da Vinci Surgical System
  Interventions: Procedure: Robotic-Assisted Radical Prostatectomy
- Laparoscopic Radical Prostatectomy (Active Comparator): Standard laparoscopic Radical Prostatectomy
  Interventions: Procedure: Laparoscopic Radical Prostatectomy

INTERVENTIONS:
Procedure: Robotic-Assisted Radical Prostatectomy
  Arms: Robotic-Assisted Radical Prostatectomy
Procedure: Laparoscopic Radical Prostatectomy
  Arms: Laparoscopic Radical Prostatectomy

SUMMARY:
In this observational cost efficacy study, the investigator compare the Laparoscopic Radical Prostatectomy (LRP) versus Robotic-Assisted Laparoscopic Prostatectomy (RALP). Every cost of care that include hospitalization related or post operative medical consumption are obtained and recorded up to 5 years follow up. Functional results (continence, potency, quality of life) are obtained through standardised questionnaires. Carcinologic results are estimated by Prostate Specific Antigen (PSA) relapse and salvage treatments. Economic evaluation will be made to estimate direct costs of the four postoperative year along with the incremental cost-effectiveness ratio (ICER) per successful surgical treatment (preserved urinary continence and erectile function and PSA < 0.2).

ELIGIBILITY:
Inclusion Criteria:

* Localized prostate cancer
* Gleason grade ≤ 3 + 4
* PSA < 15 ng / mL
* Stage ≤ T2b
* Eligible to receive laparoscopic radical prostatectomy
* Candidate bilateral or unilateral erectile preservation

Exclusion Criteria:

* Patient at high risk of postoperative progression (PSA> 15 ng / mL; grade 5 predominant, clinical or radiological stage T3
* Presenting erectile dysfunction (IIEF < 22)
* Past history of urinary incontinence (> grade 1 WHO)
* Body mass index > 30

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Erectile function | 12 months after surgery
  Proportion of patients with recovery of erectile function between T0 (before surgery) and 12 months after surgery. Recovery is defined as a maximum decrease of 5 points score of the International Index of Erectile Function (IIEF) between pre and postoperative evaluations.

SECONDARY OUTCOMES:
Surgical margins | During surgery
Prostate Specific Antigen (PSA) | Before surgery (T0), 6 months (M6), 12 months (M12), 24 months (M24) and 60 months (M60) after surgery
Continence | Before surgery (T0), 6 months (M6), 9 months (M9),12 months (M12), 24 months (M24) and 60 months (M60) after surgery
  Continence is assessed by the International Prostate Symptom Score (IPSS)
Tolerance | Perioperative period, 6 months (M6), 12 months (M12) and 24 months (M24) afer surgery
  Adverse events related to the perioperative prostatectomy, 6 months, 12 months and 24 months afer surgery
Quality of life | Before surgery (T0), 6 months (M6), 9 months (M9),12 months (M12) and 24 months (M24) after surgery
  Quality of life is assessed by EQ-5D, QLQ-C30 and QLQ-PR25 scores
Incremental cost-effectiveness ratio | 60 months afet surgery
  Economic evaluation will be made to estimate direct costs of the five postoperative years along with the incremental cost-effectiveness ratio (ICER) per successful surgical treatment

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service d'Urologie - Clinique St Augustin, Bordeaux
  - Service d'Urologie et Chirurgie de la Transplantation - Hôpital Edouard Herriot -Hospices Civils de Lyon, Lyon
  - Service d'Urologie - Institut Mutualiste Montsouris, Paris